CLINICAL TRIAL: NCT03447262
Title: A Phase 3, Open-label Study Evaluating the Long Term Safety and Efficacy of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous or Heterozygous for the F508del Mutation
Brief Title: A Study Evaluating the Long Term Safety and Efficacy of VX-659 Combination Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: At Sponsor's Discretion
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX17-659-105; 2017-004134-29 (EudraCT Number)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-659/TEZ/IVA TC (Experimental): Participants from parent studies VX17-659-102 (NCT03447249) or VX17-659-103 (NCT03460990) were administered VX-659 240 milligrams (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the TC treatment period for up to 96 weeks in the current study VX17-659-105.
  Interventions: Drug: VX-659/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: VX-659/TEZ/IVA — Fixed-dose combination tablets for oral administration qd in the morning.
  Other Names: VX-659/VX-661/VX-770; VX-659/tezacaftor/ivacaftor
Drug: IVA — IVA tablet qd in the evening.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the long-term safety and tolerability of VX-659 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous or heterozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

* Completed study drug treatment in a parent study; or had study drug interruption(s) in a parent study but completed study visits up to the last scheduled visit of the Treatment Period in the parent study.

Exclusion Criteria:

* History of drug intolerance in a parent study that would pose an additional risk to the subject in the opinion of the investigator.
* Current participation in an investigational drug trial (other than a parent study)

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (100):
- United States (48):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Medical Center, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Orlando Health, Inc.- Arnold Palmer Hospital for Children (APH), Orlando, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - Advocate Children's Hospital - Park Ridge / North Suburban Pulmonary and Critical Care Consultants, Niles, Illinois
  - Indiana Clinical Research Center, IU Health University Hospital, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Spectrum Health Medical Group Adult Cystic Fibrosis Care Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine/ St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock, Manchester, Manchester, New Hampshire
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - CF Therapeutics Development Center of Western New York, Buffalo, New York
  - Northwell Health, Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Drexel University College of Medicine / Drexel Adult Cystic Fibrosis Center, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center- Adult Cystic Fibrosis Clinic, Knoxville, Tennessee
  - Children's Foundation Research Center / Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah/ Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Pediatric Pulmonary & Cystic Fibrosis Clinic, Spokane, Washington
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne
  - Institute for Respiratory Health, Sir Charles Gairdner Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute and John Hunter Children's Hospital, New Lambton
  - Telethon Kids Institute, Perth
  - Sydney Children's Hospital, Randwick
  - Lady Cilento Children's Hospital, South Brisbane
- Canada (3):
  - Stollery Children's Hospital, Edmonton
  - Queen Elizabeth II Health Sciences Center, Halifax
  - St. Michael's Hospital, Toronto
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- Germany (9):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Clinic of J.W. Goethe University, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Mukeviszidose-Zentrum am Universitatsklinikum Jena, Klinik fuer Kinder- und Jugendmedizin, Jena
  - Universitatsklinikum Schleswig-Holstein, Klinik für Kinder- und Jugendmedizin, Lübeck
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologische Praxis Pasing, München
- Ireland (7):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Our Lady's Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Temple Street Children's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
- Israel (5):
  - Lady Davis Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Liver Unit, Haifa
  - Pediatrics Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Klinika Mukowiscydozy IMD Oddozial Chorob Pluc Szpzoz IM. Dzieci WarszaWY, Łomianki, Poland
- Spain (7):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infantil La Paz, Madrid
  - Parc Tauli Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Switzerland (2):
  - Lindenhofspital - Quartier Bleu, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (9):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Head and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshaw e Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - Wolfson Cystic Fibrosis Unit, City Campus, Nottingham
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 484 participants were enrolled from the parent studies VX17-659-102 (Study 659-102; NCT03447249) and VX17-659-103 (Study 659-103; NCT03460990). Out of which, 3 participants were enrolled but never dosed in the current study VX17-659-105 (Study 659-105). Therefore, the below results are presented for 481 participants.
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 12 years or older who participated in parent studies 659-102 or 659-103. Eligible participants from the parent studies were enrolled in the current study 659-105.
Groups:
- VX-659/TEZ/IVA Triple Combination (TC): Participants from the parent studies 659-102 or 659-103 were administered VX-659 240 milligrams (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the TC treatment period for up to 96 weeks in the current study 659-105.
Period: Overall Study
Arm/Group | VX-659/TEZ/IVA Triple Combination (TC)
Started | 481
Completed | 2
Not Completed | 479
Not completed — Adverse Event | 7
Not completed — Withdrawal of Consent (not due to AE) | 2
Not completed — Commercial Drug is Available for Participant | 9
Not completed — Death | 2
Not completed — Study Termination by Sponsor | 455
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Groups:
- VX-659/TEZ/IVA TC: Participants from parent studies 659-102 or 659-103 were administered VX-659 240 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the TC treatment period for up to 96 weeks in the current study 659-105.
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219
  Male | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 462
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 474
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to 28 Days After Last Dose of Study Drug or to the Completion of Study Participation Date, Whichever Occurs First in the Current Study 659-105 (up to Week 100)
Population: Open label safety set (OL-SS) included all participants who received at least 1 dose of study drug in the current study 659-105.
Measure: Number; unit: participants
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 481
participants
  Participants With AEs | 470
  Participants With SAEs | 99

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for Participants From the Parent Study 659-102
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: Open label full analysis set (OL-FAS) included all rolled over participants from the parent study 659-102 who received at least 1 dose of study drug in the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: percentage points
Groups:
- VX-659/TEZ/IVA TC: Participants who either received placebo (matched to VX-659/TEZ/IVA) or VX-659/TEZ/IVA in the parent study 659-102 were administered VX-659 240 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the TC treatment period for up to 96 weeks in the current study 659-105.
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 371
percentage points
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 14.2 (7.8)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 188
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 10.3 (9.3)

3. Secondary Outcome: Absolute Change in ppFEV1 for Participants From the Parent Study 659-103
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: OL-FAS included all rolled over participants from the parent study 659-103 who received at least 1 dose of study drug in the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: percentage points
Groups:
- VX-659/TEZ/IVA TC: Participants who either received TEZ/IVA or VX-659/TEZ/IVA in the parent study 659-103 were administered VX-659 240 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the TC treatment period for up to 96 weeks in the current study 659-105.
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
percentage points
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 56
  TEZ/IVA - VX-659/TEZ/IVA | 15.1 (11.9)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 54
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 11.5 (9.8)

4. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl) for Participants From the Parent Study 659-102
Description: Sweat samples were collected using an approved collection device. The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 24 (Study 659-105)
Population: OL-FAS included all rolled over participants from the parent study 659-102 who received at least 1 dose of study drug in the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 371
millimole per liter (mmol/L)
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | -48.9 (20.4)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 188
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | -49.7 (20.1)

5. Secondary Outcome: Absolute Change in SwCl for Participants From the Parent Study 659-103
Description: Sweat samples were collected using an approved collection device. The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 24 (Study 659-105)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
mmol/L
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 56
  TEZ/IVA - VX-659/TEZ/IVA | -45.7 (16.8)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 54
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | -53.5 (16.2)

6. Secondary Outcome: Number of Pulmonary Exacerbations (PEx) for Participants From the Parent Study 659-102
Description: PEx was defined as treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for at least 4 sinopulmonary signs/symptoms. The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in the parent study 659-102 or/and VX-659/TEZ/IVA in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline except for Placebo - VX-659/TEZ/IVA category, for which the baseline was defined as study 659-105 baseline.
Time Frame: From Baseline up to Week 96 (Study 659-105)
Population: The cumulative TC efficacy set for PEx analysis included all participants who were randomized to VX-659/TEZ/IVA arm and received at least one dose of study drug during the parent study 659-102 and/or received at least one dose of study drug during the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Number; unit: PEx events
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 375
PEx events
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 60
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 192
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 84

7. Secondary Outcome: Number of PEx for Participants From the Parent Study 659-103
Description: PEx was defined as treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for at least 4 sinopulmonary signs/symptoms. The analysis was planned to be reported for overall participants from the parent study 659-103, that is combined for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in the parent study 659-103 or/and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline except for TEZ/IVA - VX-659/TEZ/IVA category, for which the baseline was defined as study 659-105 baseline.
Time Frame: From Baseline up to Week 96 (Study 659-105)
Population: The cumulative TC efficacy set for PEx analysis included all participants who were randomized to VX-659/TEZ/IVA arm and received at least one dose of study drug during the parent study 659-103 and/or received at least one dose of study drug during the current study 659-105.
Measure: Number; unit: PEx events
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
PEx events | 39

8. Secondary Outcome: Number of Participants With at Least One PEx for Participants From the Parent Study 659-102
Description: PEx was defined as treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for at least 4 sinopulmonary signs/symptoms. The time-to-first-PEx data were planned to be estimated using the Kaplan-Meier (KM) method. However, because way less than 50% of participants had events, median time-to-first event data were not estimable. Instead, the number of participants with at least one PEx event was assessed and reported separately for those in Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and the VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in the parent study 659-102 or/and VX-659/TEZ/IVA in the current study 659-105). Baseline was defined as the parent study baseline except for Placebo - VX-659/TEZ/IVA category, for which the baseline was defined as study 659-105 baseline.
Time Frame: From Baseline up to Week 96 (Study 659-105)
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- VX-659/TEZ/IVA TC: Participants who either received placebo (matched to VX-659/TEZ/IVA), TEZ/IVA or VX-659/TEZ/IVA in the parent studies 659-102 or 659-103 were administered VX-659 240 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the TC treatment period for up to 96 weeks in the current study 659-105.
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 375
participants
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 43
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 192
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 52

9. Secondary Outcome: Number of Participants With at Least One PEx for Participants From the Parent Study 659-103
Description: PEx was defined as treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for at least 4 sinopulmonary signs/symptoms. The time-to-first-PEx data were planned to be estimated using the KM method. However, because way less than 50% of participants had events, median time-to-first-event data were not estimable. Instead, the number of participants with at least one PEx event was assessed and reported for all participants from the parent study 659-103, that is combined for those in the TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and the VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in the parent study 659-103 or/and in the current study 659-105). Baseline was defined as the parent study baseline except for TEZ/IVA - VX-659/TEZ/IVA category, for which the baseline was defined as study 659-105 baseline.
Time Frame: From Baseline up to Week 96 (Study 659-105)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
participants | 28

10. Secondary Outcome: Absolute Change in Body Mass Index (BMI) for Participants From the Parent Study 659-102
Description: BMI was defined as weight in kilograms (kg) divided by squared height in meters (m^2). The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 371
kilogram per meter square (kg/m^2)
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 1.55 (1.35)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 188
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 1.43 (1.94)

11. Secondary Outcome: Absolute Change in BMI for Participants From the Parent Study 659-103
Description: BMI was defined as weight in kg divided by squared height in meters (m^2). The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
kg/m^2
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 56
  TEZ/IVA - VX-659/TEZ/IVA | 1.16 (1.68)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 54
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 0.90 (1.52)

12. Secondary Outcome: Absolute Change in BMI Z-score for Participants From the Parent Study 659-102 (Participants <=20 Years Old at Parent Study Baseline)
Description: BMI was defined as weight in kg divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard. The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 60 (Study 659-105)
Population: OL-FAS included all rolled over participants from the parent study 659-102 who were <=20 years old at parent study baseline and received at least 1 dose of study drug in the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 114
z-score
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 57
  Placebo - VX-659/TEZ/IVA | 0.22 (0.59)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 57
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 0.10 (0.44)

13. Secondary Outcome: Absolute Change in BMI Z-score for Participants From The Parent Study 659-103 (Participants <=20 Years Old at Parent Study Baseline)
Description: BMI was defined as weight in kg divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard. The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 60 (Study 659-105)
Population: OL-FAS included all rolled over participants from the parent study 659-103 who were <=20 years old at parent study baseline and received at least 1 dose of study drug in the current study 659-105. Here, "number analyzed" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 30
z-score
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 16
  TEZ/IVA - VX-659/TEZ/IVA | NA (NA) — As pre-specified in analysis plan, due to less than 20 number of participants in the TEZ/IVA - VX-659/TEZ/IVA category, the summary statistics were no longer applicable. Therefore, no BMI z-score efficacy data is available for this category.
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 14
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | NA (NA) — As pre-specified in analysis plan, due to less than 20 number of participants in the VX-659/TEZ/IVA - VX-659/TEZ/IVA category, the summary statistics were no longer applicable. Therefore, no BMI z-score efficacy data is available for this category.

14. Secondary Outcome: Absolute Change in Body Weight for Participants From the Parent Study 659-102
Description: The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 371
kg
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 4.8 (4.4)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 188
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 4.3 (5.6)

15. Secondary Outcome: Absolute Change in Body Weight for Participants From the Parent Study 659-103
Description: The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
kg
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 56
  TEZ/IVA - VX-659/TEZ/IVA | 3.7 (4.9)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 54
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 3.2 (5.0)

16. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for Participants From the Parent Study 659-102
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. The analysis was planned to be reported separately for Placebo - VX-659/TEZ/IVA category (participants who received placebo in the parent study 659-102 and VX-659/TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-102 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 371
units on a scale
  Placebo - VX-659/TEZ/IVA: number analyzed (Participants) | 183
  Placebo - VX-659/TEZ/IVA | 16.7 (18.7)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 188
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 19.7 (17.4)

17. Secondary Outcome: Absolute Change in CFQ-R Respiratory Domain Score for Participants From the Parent Study 659-103
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. The analysis was planned to be reported separately for TEZ/IVA - VX-659/TEZ/IVA category (participants who received TEZ/IVA in the parent study 659-103 and VX-659-TEZ/IVA in the current study 659-105) and VX-659/TEZ/IVA - VX-659/TEZ/IVA category (participants who received VX-659/TEZ/IVA in both the parent study 659-103 and in the current study 659-105) as pre-specified in analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Week 72 (Study 659-105)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 110
units on a scale
  TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 56
  TEZ/IVA - VX-659/TEZ/IVA | 17.1 (18.2)
  VX-659/TEZ/IVA - VX-659/TEZ/IVA: number analyzed (Participants) | 54
  VX-659/TEZ/IVA - VX-659/TEZ/IVA | 16.9 (17.3)

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days After Last Dose of Study Drug or to the Completion of Study Participation Date, Whichever Occurs First in the Current Study 659-105 (up to Week 100)
Arm/Group | VX-659/TEZ/IVA TC
All-Cause Mortality (participants affected / at risk) | 2/481
Serious Adverse Events (participants affected / at risk) | 99/481
Other Adverse Events (participants affected / at risk) | 446/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-659/TEZ/IVA TC (N=481)
Cardiac failure acute (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 6
Duodenitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Generalised oedema (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 40
Influenza (Infections and infestations) | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Medical device site cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia pseudomonal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Stoma site extravasation (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood creatine phosphokinase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Pulmonary function test decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Device leakage (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Breathing-related sleep disorder (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-659/TEZ/IVA TC (N=481)
Abdominal pain (Gastrointestinal disorders) | 42
Abdominal pain upper (Gastrointestinal disorders) | 26
Diarrhoea (Gastrointestinal disorders) | 42
Nausea (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 27
Fatigue (General disorders) | 31
Pyrexia (General disorders) | 56
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 149
Influenza (Infections and infestations) | 40
Nasopharyngitis (Infections and infestations) | 97
Sinusitis (Infections and infestations) | 30
Upper respiratory tract infection (Infections and infestations) | 104
Viral upper respiratory tract infection (Infections and infestations) | 38
Alanine aminotransferase increased (Investigations) | 43
Aspartate aminotransferase increased (Investigations) | 42
Blood creatine phosphokinase increased (Investigations) | 37
Headache (Nervous system disorders) | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 126
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 39
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 53
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 80
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 28
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 40
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 27
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 69
Rash (Skin and subcutaneous tissue disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03447262/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT03447262/SAP_001.pdf